CLINICAL TRIAL: NCT05956717
Title: The Effect of Orthokeratography on the Quality of Life and Behavior of Myopic Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023032
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental Group: Subjects wore orthokeratology lenses
  Interventions: Device: Orthokeratology
- Control group: Subjects wore single-vision glasses group

INTERVENTIONS:
Device: Orthokeratology — The experimental group wore orthokeratology lenses
  Groups: Experimental Group

SUMMARY:
The study intended to observe the changes in the quality of life, behavior, and eye habits of children and adolescents aged 8-18 years before and after orthokeratology, as well as the differences in the quality of life and behaviors of different myopic groups after keratoplasty, using the EQ-5D-Y, CHU9D, and CHROME-G scales with the use of a self-assessment method.

ELIGIBILITY:
Inclusion Criteria:

* Spherical equivalent ranged -1.00D from-5.00D
* Optimal corrected visual acuity ≥1.0 in both eyes
* No apparent strabismus or other eye disease
* Able to read Chinese and communicate in Mandarin, able to understand the questions in the questionnaire

Exclusion Criteria:

* A history of corneal surgery within 1 year
* Eyelid abnormalities or infection
* An inability to wear orthokeratology
* Use medications that affect the wear of eye and corneal contact lenses
* Those who have participated in a clinical trial of a drug within 90 days
* Allergic patients who have used contact lenses and/or care products
* The researchers consider it inappropriate to participate in this program

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents aged 8-18 years with normal eye health
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in EuroQol five dimensions questionnaire(EQ-5D-Y) score | The change was the difference between each two follow-up times, including before and one day, one week, one month and three months after orthokeratology
  The health utility can be calculated by the number of the answer to the question. 0 means death and 1means complete health.
Changes in the Child Health Utility 9D (CHU9D) score | The change was the difference between each two follow-up times, including before and one day, one week, one month and three months after orthokeratology
  The health utility can be calculated by the number of the answer to the question. 0 means death and 1means complete health.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, China